CLINICAL TRIAL: NCT06670261
Title: JUNE Project: Does the Modeling of Nasal Airflows Improve the Pathophysiological Understanding and the Diagnosis of Functional Respiratory Disorders?
Brief Title: Diagnosis of Respiratory Disorders by the Numerical Modeling.
Acronym: JUNE
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: CREATIS Laboratory (Unknown); Optifluides (Unknown)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2023/62
Record Dates: First submitted 2024-10-30; First posted 2024-11-01 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Nasal Obstruction; Deviated Nasal Septum
Keywords: Numerical modeling; Fluid Dynamics; Computer simulation; Septoplasty; Nasal Air Flow; Sinonasal CT-Scan; Computational Fluid Dynamic Simulation
MeSH Terms: conditions — Nasal Obstruction | interventions — Data Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy subjects: 100 patients without ONC
  Interventions: Other: Data collection
- Patients with CNO: 200 patients with anatomical ONC
  Interventions: Other: Data collection

INTERVENTIONS:
Other: Data collection — Retrospective pseudo-anonymized clinical and scannographic data from the routine management of patients in rhino-sinusology consultations.

SUMMARY:
Chronic Nasal obstruction (CNO) is not currently measurable objectively because clinicians use validated declarative self-questionnaires whose results are linked to the level of understanding, the acute or chronic clinical situation, fatigue, psychological state and the desired gain. Using numerical simulations of the passage of air in the nasal cavities determining specific airflow parameters, the respiratory comfort of healthy subjects and the CNO of patients treated for this pathology could be explained.

DETAILED DESCRIPTION:
CNO concerns 20 to 25% of the general population due to numerous etiologies (septal deviation, polyps, chronic rhinosinusitis, post-therapeutic cancer quality of life…). It disrupts sleep and deteriorates all the compartments of the quality of life sometimes to depression. To date, nobody knows the exact component of CNO which is probably the amalgamation of different mucosal information and all measurement attempts have failed by lack of reliability and reproducibility. This major shortcoming of CNO quantification leads to diagnosis uncertainties, quantification of symptoms and therapeutic. The place of such complementary exam able to do an objective measure of NO is expected by the profession. The Computational Fluid Dynamic Simulation (CDFS) of the air passage would allow a complementary functional analysis to anatomy of the sino-nasal cavities to measure CNO. Such information would reduce the failure rate and unnecessary functional surgeries by 25%, reduce the inappropriate care of patients suffering to obstructive sleep disorders and reduce the financial burden on the health system. No patient follow-up in this study: pseudo-anonymized retrospective clinical and scannographic data from the routine management of patients in rhinosinusology consultations.

ELIGIBILITY:
Inclusion Criteria:

* 18 years ≤ age < 70 years
* BMI < 30 kg/m2
* Subject or Patient of Caucasian ethnic origin or from the Mediterranean region.
* Asymptomatic subject with or without a septal deviation without sinonasal disease with a NOSE score ≤ 7 Or Patient suffering from chronic nasal obstruction of morphological origin (symptomatic septal or nasoseptal deviation) requiring surgical management with a NOSE score ≥ 9/20, without or .with sleep apnea with an Apnea-hypopnea index ≤ 20 with no other cause than this apnea syndrome

Exclusion Criteria:

* Acute or chronic rhinosinusitis with or without polyps (except controlled allergic rhinitis)
* Vasculitis
* Empty nasal cavity syndrome
* Septal perforations
* History of nasal plastic surgery, sinonasal endoscopic surgery and cancer with head or neck radiotherapy
* Uncontrolled bronchopulmonary pathology
* Treatments with nasal vasomotor repercussions.

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: participant with or without chronic nasal obstruction seen in the rhinology department of Bordeaux University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-07-09 (Actual); Primary Completion 2026-07-09 (Estimated); Study Completion 2026-07-09 (Estimated)

PRIMARY OUTCOMES:
Correlation coefficient | at inclusion (day 0)
  Correlation coefficient of at least one of the simulation parameters greater than 0.5 with the NOSE score in a healthy population and a pathological population. This parameter could be Pressure (P), Temperature (T), mass exchanges (C) and/or shear stresses (SS).

SECONDARY OUTCOMES:
Physical values of air flow | at inclusion (day 0)
  Physical values of air flow in the normal population and in the pathological population suffering from ONC, during resting breathing for all CFD parameters at 0.5 sec from the start of the respiratory cycle.
flow parameters | at inclusion (day 0)
  Statistical comparison of the flow parameters between these two groups and correlation of clinical data with the flow parameters.
weighting coefficients of the flow parameters | at inclusion (day 0)
  Search for the weighting coefficients of the flow parameters and validation of the equation determining the CNO.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Bordeaux, Bordeaux, France

IPD SHARING:
Plan to Share IPD: Undecided